CLINICAL TRIAL: NCT05574920
Title: Accuracy and Safety of Al18F-NOTA-FAPI-04 PET/CT in the Diagnosis of Axillary Lymph Node Metastasis in Early Breast Cancer Patients: A Prospective Cohort Study
Brief Title: Characterizing Breast Cancer With Al18F-NOTA-FAPI-04 PET/CT (PFB-02)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-FAPI-BC-2
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-FAPI-04 PET/CT (Experimental): Inject Al18F-NOTA-FAPI-04 and then perform PET/CT scan.
  Interventions: Diagnostic Test: Al18F-NOTA-FAPI-04 PET/CT scan

INTERVENTIONS:
Diagnostic Test: Al18F-NOTA-FAPI-04 PET/CT scan — Patients enrolled underwent PET/CT after injection of Al18F-NOTA-FAPI-04 to image lesions of breast cancer.

SUMMARY:
Fibroblast activation protein (FAP) is overexpressed in cancer-associated fibroblasts (CAFs), which constitute a major proportion of cells within the tumor microenvironment, especially in breast cancer. Previous studies have demonstrated that FAPI PET/CT performs well in cases of epithelial tumors, including breast cancer. This prospective study is going to investigate the performance and value of Al18F-NOTA-FAPI-04 PET/CT in patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a complex, heterogeneous disease comprising numerous distinct biological subtypes characterized by variant pathobiological features and clinical behaviors. 18F-fluorodeoxyglucose (18F-FDG) PET/CT, an essential imaging modality in the characterization of metabolism within the tumor, has successfully evolved in the diagnosis, staging, and assessment of treatment response in patients with breast cancer. Cancer-associated fibroblasts (CAFs) are a crucial component of the tumor stroma with diverse functions. Fibroblast activation protein (FAP), a type II membrane-bound glycoprotein from the dipeptidyl peptidase-4 family, is highly expressed in the CAFs of several epithelial carcinomas, including breast cancer, coupled with relatively low expression in normal tissue. Based on this characteristic, many small-molecule inhibitors of FAP (FAPIs) labeled with radioactive tracers (68Ga, 18F, or 177Lu) have been synthesized as theranostic radiotracers for cancer. Previous studies on FAPI PET/CT tumor imaging have focused on the 68Ga radionuclide rather than 18F. As 18F-labeled FAPI has more favorable physical properties, high production capacity, and good imaging characteristics, it may be an ideal agent for PET imaging. Therefore, this study aims to evaluate the performance and value of Al18F-NOTA-FAPI-04 PET/CT in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old;
* newly diagnosed BC confirmed by biopsy or with BI-RADS category 4C or 5 lesions by US or MG;
* BC clinical stagecT1-3 cN0-3 M0;
* no prior treatment for BC.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* patients who were unwilling to undergo PET/CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance (1) | Through study completion, an average of 1 year
  Diagnostic performance including sensitivity, specificity, accuracy, positive predictive value and negative predictive value of Al18F-NOTA-FAPI-04 PET/CT in the detection of ALN metastasis according to the pathological reference standard on a per-patient basis, compared with 18F-FDG PET/CT and ultrasound.

SECONDARY OUTCOMES:
Clinical Stage | Through study completion, an average of 1 year
  Clinical stage changed by Al18F-NOTA-FAPI-04 PET/CT compared to 18F-FDG PET/CT.
Diagnostic Performance (2) | Through study completion, an average of 1 year
  Diagnostic performance of ALN metastasis of Al18F-NOTA-FAPI-04 PET/CT with or without previous biopsy on breast lesion.
Safety | Through study completion, an average of 1 year
  Short-term adverse effects (AEs) after Al18F-NOTA-FAPI-04 injection.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China